CLINICAL TRIAL: NCT05762094
Title: A Retrospective Study on Personalized Dosing Strategy of Patients With Bacterial Infections Treated by Carbapenems From a Tertiary Medical Center During 2018-2021
Brief Title: A Retrospective Study on Personalized Dosing Strategy of Patients Treated by Carbapenems: 2018-2021
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-504-01
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-02

CONDITIONS: Bacterial Infections
Keywords: Carbapenem; Bacterial Infections
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CAR-R: Patients with impaired renal function (eGFR < 60ml/min/1.73m2) treated by carbapenem
- CAR-L: Patients with liver cirrhosis or impaired liver function (Child-Pugh grade B or C) treated by carbapenem
- CAR-LR: Patients with co-morbidity of both liver cirrhosis or impaired liver function (Child-Pugh grade B or C) and impaired renal function (eGFR < 60ml/min/1.73m2) treated by carbapenem
- CAR-N: Patients with normal liver function or renal function treated by carbapenem

SUMMARY:
Patients may benefit from the personalized carbapenem dosing strategy based on pharmacokinetics. The objective of this study is to retrospectively review and analyze the clinical outcomes of patients with different dosing strategy.

DETAILED DESCRIPTION:
Rational use of carbapenem is closely associated with the clinical outcome of patients with infections. Serum concentration of carbapenem varies from different populations. The objective of this study is to describe the clinical outcome of patients with infection treated by carbapenem in China, regarding diagnosis, treatment and follow-up. It is a single-center, retrospective, descriptive study. Inclusion criteria are an age ≥ 18, diagnosed as bacteria infection and serum concentration must be determined during therapy. Data concerning clinical presentation, biological samples, treatment and follow-up will be assessed. A descriptive analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

Age over 18 years Chinese patient: male or female Diagnosed as bacterial infection Treated by carbapenem Serum concentration determined during therapy

Exclusion Criteria:

Duration of carbapenem treatment less than 48 hours Patients renal or liver function not tested before treatment started Using more than two kinds of carbapenem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese adult patients with bacterial infections treated by carbapenem
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | January 2018-December 2021
  30-day mortality and 90-day mortality
Attainment of Target Trough Concentration | January 2018-December 2021
  Attainment of Target Trough Concentration

SECONDARY OUTCOMES:
Proportion of patients reach clinical response at end of treatment | January 2018-December 2021
  By definition, a successful clinical response means resolution of clinically significant signs and symptoms(defined as any criteria of systemic inflammatory response syndrome, body temperature over 38℃ or below 36℃, blood white cell count more than 12*10^9/L or less than 4*10^9/L, respiratory rate faster than 20 times per minute and heart rate higher than 90 beats per minute) or partial resolution of clinically significant signs and symptoms
Proportion of patients reach clinical response at day 4 of treatment | January 2018-December 2021
  By definition, a successful clinical response means resolution of clinically significant signs and symptoms(defined as any criteria of systemic inflammatory response syndrome, body temperature over 38℃ or below 36℃, blood white cell count more than 12*10^9/L or less than 4*10^9/L, respiratory rate faster than 20 times per minute and heart rate higher than 90 beats per minute) or partial resolution of clinically significant signs and symptoms
Daily Sequential Organ Failure Assessment score change | January 2018-December 2021
  Sequential Organ Failure Assessment score (Range from 0-24), lower score means a better outcome. Increase of 2 points within 48 hours means the presence of sepsis.
Incidence of Septic Shock | January 2018-December 2021
  Incidence of Septic Shock
Safety outcome measures | January 2018-December 2021
  Safety outcome measures including nephrotoxicity, hepatotoxicity and other adverse events related to the antibiotic treatment of carbapenems

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided